CLINICAL TRIAL: NCT05823220
Title: A Pragmatic Randomized Trial Integrating Homelessness Diversion Services Into an Emergency Department Discharge System
Brief Title: A Pragmatic Trial Integrating Homelessness Diversion Services Into an Emergency Department Discharge System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jack Tsai, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-SPH-22-0762; R01MD018213 (NIH)
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Homelessness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homeless diversion (HD) group (Experimental)
  Interventions: Behavioral: Homeless diversion (HD)
- Treatment-as-usual (TAU) group (Active Comparator)
  Interventions: Behavioral: Treatment-as-usual (TAU)

INTERVENTIONS:
Behavioral: Homeless diversion (HD) — Participants will receive services from specialty-trained community health workers and will be invited to complete monthly assessments via text and phone to assess their health and housing for 6 months and to share feedback on their experience with the intervention after completion by a text message to a link for the survey
  Arms: Homeless diversion (HD) group
Behavioral: Treatment-as-usual (TAU) — Participants will receive a list of community resources they can contact to receive services and will be invited to complete monthly assessments via text and phone to assess their health and housing for 6 months and to share feedback on their experience with the intervention after completion by a text message to a link for the survey
  Arms: Treatment-as-usual (TAU) group

SUMMARY:
The purpose of this study is to determine whether a homelessness diversion program integrated into a hospital emergency department (ED) will lower ED use, to identify characteristics of individuals most likely to benefit from homelessness diversion and to discover opportunities to tailor Homelessness Diversion (HD) services to better meet the needs of diverse communities.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* discharged from a Harris Health Hospital ED (Ben Taub or LBJ)
* at imminent risk of homelessness
* patients with Medicaid, Medicare or who are uninsured

Exclusion Criteria:

* having a conservator (legal guardian)
* plans to move away from Texas in 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of ED visits | end of study (6 months after start of study)

SECONDARY OUTCOMES:
Number of participants who experience homelessness | end of study (6 months after start of study)
Change in health related quality of life as assessed by the Short Form-12 version 2.0 (SF12v2) health Survey | baseline, month 1, month 2, month 3, month 4, month 5 and month 6
  This is a 12 item questionnaire and scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Tsai, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No